CLINICAL TRIAL: NCT02402270
Title: An Adaptive, Single-Blind, Parallel, Randomized, Phase 2, Formulation Screening/Proof of Concept, Safety, Tolerability and Efficacy Study of Three Formulations/Dosing Regimens of ECP (PEG 3350) Colon Prep Kit Compared to Comparators.
Brief Title: Safety and Tolerability Study of an Edible Colon Preparation
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: ColonaryConcepts LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: ECP-002
Record Dates: First submitted 2015-03-25; First posted 2015-03-30 (Estimated); Last update posted 2018-01-29 (Actual); Status verified 2018-01

CONDITIONS: Bowel Preparation
Keywords: Colonoscopy; Preparation
MeSH Terms: interventions — polyethylene glycol 3350; MoviPrep

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (5):
- ECP-019 A (Group A) (Experimental)
  Interventions: Drug: ECP-019
- ECP-019 B (Group B) (Experimental)
  Interventions: Drug: ECP-019
- ECP-019 C (Group C) (Experimental)
  Interventions: Drug: ECP-019
- Group D (Active Comparator)
  Interventions: Drug: MoviPrep® (PEG 3350)
- Group E (Active Comparator)
  Interventions: Drug: NuLYTELY® (PEG 3350)

INTERVENTIONS:
Drug: NuLYTELY® (PEG 3350)
  Arms: Group E
Drug: ECP-019
  Arms: ECP-019 A (Group A); ECP-019 B (Group B); ECP-019 C (Group C)
Drug: MoviPrep® (PEG 3350)
  Arms: Group D

SUMMARY:
The purpose of this study is to learn about a new bowel preparation that uses food to clean the colon.

In order to learn about this new food preparation, some people in this study will get the food preparation, and others will get the standard liquid bowel preparation.

Patients will be randomized (like flipping a coin) to one of five groups:

Group 1 - Menu A Meal Kit - contains bars, shakes, soup, and a rice bowl Group 2 - Menu B Meal Kit - contains bars, shakes, soup, and a rice bowl Group 3 - Menu C Meal Kit - contains bars and shakes Group 4 - MoviPrep Group 5 - NuLYTELY

DETAILED DESCRIPTION:
The purpose of this Phase 2 formulation screening/proof of concept study is to evaluate the safety, tolerability, and efficacy of up to 3 ECP-019 formulations/dosing regimens comprising a PEG 3350 Colon Prep Kit, containing electrolytes provided by the foods, in 3 formulations/ dosing regimens as compared to 2 comparators in a Phase 2 study.

ELIGIBILITY:
Inclusion Criteria:

* Patients whose physician has prescribed colonoscopy for colorectal cancer screening or surveillance for colorectal cancer.
* Patients with a previous history of completing a bowel cleansing procedure for a colonoscopy.

Exclusion Criteria:

* Known intestinal stricture of any etiology.
* History of diabetes mellitus.

Ages: 18 Years to 74 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 69 (Actual)
Dates: Start 2015-05 (Actual); Primary Completion 2016-06 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
The proportion of patients with successful colon cleansing as assessed by the blinded gastroenterologists using the Aronchick Scale. | One year

SECONDARY OUTCOMES:
Percentage of patients who completed each of the ECP-019 formulation/dosing regimens | One year

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Indianapolis, Indiana
  - Lebanon, New Hampshire